CLINICAL TRIAL: NCT04826029
Title: Randomized Study Evaluating the Impact on the Cost and Quality of Life of Follow up by Systematic Imaging in Patients With Advanced Stage Ovarian, Fallopian Tube or Primary Peritoneum Cancer
Brief Title: Impact of Systematic Imaging for Follow up of Patients With Ovarian, Fallopian Tube or Primary Peritoneum Cancer
Acronym: QUALOV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer feasible because of new recommendations (RPC St Paul de Vence) which advocate the performance of systematic imaging in addition to CA 125 in patients treated in first line maintenance in order not to ignore a relapse (2021).
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP200051; 2020-A02836-33 (Other: ANSM)
Record Dates: First submitted 2021-03-08; First posted 2021-04-01 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Advanced Stage Serous Epithelial Cancer of the Ovary; Advanced Stage Cancer of Tubes; Advanced Stage Cancer of Peritoneum
Keywords: Ovarian cancer; Recurrence; Imaging follow up; HE4; CA125
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (Other)
  Interventions: Other: Standard strategy
- Interventional arm (Experimental)
  Interventions: Other: Follow-up strategy

INTERVENTIONS:
Other: Standard strategy — In the standard arm, patients will complete CA 125 (+/- HE4) at 3 months, 6 months, 12 months, 18 months and 24 months (+/- 15 days), complete the HAD and EQ5D self-questionnaires, and be managed according to INCa 2018 recommendations. If clinical symptoms, marker elevation, and/or imaging workup occur, the patient will be referred to the multidisciplinary consultation meeting (MDC) for management according to INCa 2018.
  Arms: Standard arm
Other: Follow-up strategy — In the interventional arm, patients will perform at 3 months, 6 months, 12 months, 18 months and 24 months (+/- 15 days) a CA125 assay (+/- HE4 assay), a thoracoabdominal CT scan after contrast injection and a whole body MRI (T2, DW and T1 sequences after fat saturation before and after gadolinium injection) with a maximum delay of 15 days between the two examinations, and will complete the HAD and EQ5D self-questionnaires. A senior radiologist from each center will perform a prospective reading of each of the images. For any suspicious anomaly identified, the following criteria will be analyzed: Size, location, number, evolution, contrast after injection, MRI signal (T2, Diffusion, Dynamic Enhancement Curve). The RECIST criteria (version 1.1) will be applied.
  Arms: Interventional arm

SUMMARY:
After well-conducted treatment of ovarian, tubal and primary peritoneum cancer by maximum tumor reduction surgery and chemotherapy including platinum salt and paclitaxel, the clinical remission rate is over 50%. However, 75-80% of patients with ovarian, tube or primary peritoneum cancer recur within 2 years of the end of treatment. In the latest INCa recommendations for 2018, systematic imaging (thoraco-abdomino-pelvic scanner (CT), MRI, PET CT) is not recommended based on the literature because of its low added value compared to CA 125 dosage (sensitivity ranging from 67% to 95%, and specificity of 87% to 93%), its irradiating character (CT) and its cost. However, the recommendations are based on imaging studies dating back at least a decade. Since these studies, technological advances have improved the diagnostic performance of imaging: sensitivity is 78% for whole-body CT scans and 98% for full-body MRI for the diagnosis of ovarian cancer recurrence. Furthermore, previous randomized studies showed no survival benefit with early treatment of relapse on the basis of a high concentration of CA125 alone, so the value of routine CA125 measurement in the follow-up of ovarian cancer patients may be limited. These recent studies lead to heterogeneity in surveillance protocols for ovarian cancer patients despite recommendations. In addition, treatments for recurrences have evolved as well as maintenance treatments to become chronic treatments, with the emergence of the maintenance new treatments detecting early recurrence is particularly important (notably through the development of new molecules given in maintenance treatment). But early detection have to be balanced with the quality of life of these patients.

In usual care, imaging surveillance is often carried out despite the absence of recommendations or data from the literature of high level of evidence.

The question arises as to whether radiological monitoring could make an impact on patient survival without being a source of excessive false positives, patient stress and non-productive costs.

QUALOV trial is a multicenter randomized study for patients in remission after treatment of advanced stage serous epithelial ovarian, fallopian tube or primary peritoneum cancer (stage III and beyond).

The main objective is to assess the effectiveness of systematic imaging for patients followed after advanced stage serous epithelial ovarian, fallopian tube or primary peritoneum cancer

DETAILED DESCRIPTION:
This is a randomized multi-center study. Randomization will be stratified on two major prognostic factors:

* The BRCA mutation (germline or somatic)
* the serous high or low grade histological subtype of histological se topical (defined according to morphological-well-differentiated criteria, low to moderate atypia, <3-4 mitoses/10 fields-and immunohistochemical-RO - strong p16/p53 low) At J0, after obtaining informed consent or within 7 days, patients will be randomized in one of the two arms (intervention group/standard group).

In the intervention arm, patients will perform a ca125 dosing ,/he4 dosage, a thoraco abdomino pelvic CT scan after contrast product injection and a full-body MRI (T2, DW and T1 sequences after fat saturation before and after gadolinium injection) with a maximum of 15 days between the two examinations, and will complete the HAD and EQ5D self-tests. A senior radiologist from each center will perform a prospective reading of each of the imaging. For any suspicious anomaly identified, the following criteria will be analyzed: Size, location, number, scalability, contrast taking after injection, MRI signal (T2, Diffusion, Dynamic Enhancement Curve). The RECIST criteria (version 1.1) will be applied.

In the standard arm, patients will perform a dosage of CA 125 (HE4 dosage), complete the HAD and EQ5D self-questionnaires, and the patient will be managed according to the INCa 2018 recommendations.

In the case of clinical abnormality (symptoms such as pain, transit changes, increased abdominal volume; or abnormality in clinical examination such as palpation of a mass, carcinosis nodule or suspicious adenopathy), marker elevation (CA125 >2N and/or 70 IU/L, HE4 > 140 pmol/L) and/or imaging (read by a senior at the center), the patient will be referred to the Multidisciplinary Consultation Meeting (PCR) for management according to the INCa 2018 recommendations.

In the case of a biopsy or surgery recommendation, it will be performed within a maximum of 2 months (according to the recommendations of good practice).

In common practice, the diagnosis of recurrence is often based on obvious imaging elements (RECIST criteria) without histological evidence. It is only in uncertain cases that a biopsy will be performed or a diagnostic surgery, so in this study it will be placed as in current practice without adding procedures that are not performed in common practice to start a new treatment.

In terms of the management of recidivism, this is the most complex element because it is difficult to homogenize all attitudes. Indeed, many studies are still underway to define the best ways to manage recurrences with contradictory results (such as DESKTOP III in favour of new complete secondary surgery and the study by Coleman et al published in the NEJM in 11/2019 which does not find this advantage). The purpose of this study is not to be not to define (or impose) optimal support (which has yet to be defined). In addition, this study is in real life and the modalities of care can change over the duration of the study.

We will therefore follow the main standard principles of the management of recidivism based on the characterization of platinosensitivity according to recurrence at less than 6 months, 6 to 12 months or more than 12 months of recidivism. Surgery will be considered if it is a localized recurrence, accessible for complete resection and less than 6 months delay compared to the last platinum chemotherapy (use of the AGO score).

Cost-utility analysis and AIB The economic assessment will be conducted in accordance with the recommendations of the HAS (updated) and the CHEERS collaboration, by measuring prospectively on the population study population the costs and outcomes at 24 months and extrapolating them over a lifetime.

We will carry out a cost utility study, based on the measurement of survival and quality of life from the EQ 5D. We will estimate a cost-utility incremental ratio and conduct a probabilistic sensitivity analysis to locate the systematic imaging surveillance strategy at cost-effectiveness.

For the economic assessment, we selected two perspectives, the collective perspective and the perspective of Medicare. The measurement of route efficiency will be based on an analysis of the different costs from a community perspective and an analysis of clinical effectiveness in real life and will be supplemented by a budgetary impact analysis from the perspective of Medicare. The time horizon for the main study ranges from inclusion to 2 years with secondary modelling over the whole life, with an annual discount of costs and benefits at 4% for the first 30 years, 1.5% then according to the latest recommendations of the HAS.

The data will be analyzed for all patients included in the study, based on the principle of the intention-to-treat analysis. We plan to perform sub-analyses based on BRCA (germinal or somatic) stratification and histological serous subtype.

The reference intervention is the usual management of patients with a dosage of CA 125 (OR/- dosage of HE4) and management according to the INCa 2018 recommendations according to the results. The procedure studied is also a dosage of CA125 (HE4 dosage), followed by a thoraco abdominopelvic CT scan after contrast product injection and a whole body MRI. Management will be decided on the basis of the results of the examinations

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years.
* Patients in remission from proven stage III and above serous epithelial cancer of the ovary, peritoneum or tubes with complete macroscopic surgical resection (whether initial or interval)
* Signature of informed consent by the patient
* Affiliation to a French social security scheme (excluding AME)

Exclusion Criteria:

* Patients with a contraindication to MRI or CT examination (wearing a material with magnetic properties : pacemaker, ferromagnetic material, etc.)
* Intolerance to iodinated contrast or gadolinium or severe renal failure (DFG <30 ml/min/1.73 m2)
* Patients deprived of their liberty and patients Under legal protection (under guardianship or under curatorship)
* Patients participating in another interventional research (in particular research with radiological exposure as well

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
24-month incremental cost-to-utility ratio | At 24 months after inclusion
  Incremental cost-utility ratio defined as the difference in total cost at 2 years between the systematic imaging strategy and the standard strategy, relative to the difference in survival and quality of life (QALYs).

SECONDARY OUTCOMES:
Duration without treatment | At 24 months after randomization
  Duration without treatment is defined as the time between randomization at the end of the initial treatment and initiation of the following treatment (surgery or chimiotherapy)
Mean score of HAD (Hospital Anxiety and Depression scale) | at 3 months, 6 months, 12 months, 18 months and 24 months after randomization
  Hospital Anxiety and Depression scale will be used
Mean score of Quality of Life | at 3 months, 6 months, 12 months, 18 months and 24 months after randomization
  Quality of life of patients will be measured using the EQ5D questionnaire
Overall survival | At 24 months after randomization
  Overall survival is defined as the time from the date of randomization to death regardless of the cause of death.
Tumor board's decision to treat the patient for recurrence | At 24 months after randomization
  Tumor board decision elements (CA125 elevation alone, CA125 elevation and suspicious imaging, normal but normal CA125 mass detection, modification of several biological dosages, change in suspicious volume to imaging,...) will be collected and linked to
Rate of complete secondary surgery | At 24 months after inclusion
  To predict the possibility of complete resection of recurrence by surgery
Rate of surgery for recurrence | At 24 months after inclusion
  To compare the percentage of operable patients in each group
Change in caregiver preference on ideal monitoring modalities | at randomization and at 24 month after the last patient randomization (end of the study)
  Caregiver preference questions on ideal monitoring modalities :
  - "How important is imaging to you in the monitoring of ovarian, tube and primary peritoneal cancers" rated on a scale of 0 to 4.
Patient preference on ideal monitoring modalities for patient of interventional group | at 24 month after randomization
  Patient preference questions on ideal monitoring modalities :
  - "Do you think the constraints of routine follow-up imaging are acceptable for a situation like yours? " rated on a scale of 0 to 4.
Diagnostic performance of HE4 | At 24 months after inclusion
  Diagnostic performance (sensitivity, specificity, positive predictive value, negative predictive value) of CA125 and CA125-HE4 will be estimated on the subgroup of patients who had both dosages during their follow-up.
Cost/life-year gained over lifetime horizon | 2 years
  Survival measured by the area between the two Kaplan Meier curves, costs are in euros
Number of subjects to be screened to gain one | 2 years
  Number of subjects to be screened to gain one
Incremental cost-to-utility ratio | 2 years
  Incremental cost-utility ratio defined as the difference in total cost between the systematic imaging strategy and the standard strategy, relative to the difference in survival and quality of life (QALYs).
Budgetary impact at 5 years | At 5 years
  Costs in euros
Cost/complete resection of recurrent disease | At 24 months
  Cost/complete resection of recurrent disease

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Uzan, Pr, Principal Investigator — Hôpital Pitié Salpêtrière - Assitance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France